CLINICAL TRIAL: NCT04296188
Title: Comparison of Erector Spina Plane Block and Serratus Anterior Plane Block in Patients Undergoing Mastectomy
Brief Title: Erector Spina Plane Block vs Serratus Anterior Plane Block for Postoperative Mastectomy Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Mehtap Gürler Balta, asist.prof., Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19KAEK253
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Mastectomy; Pain, Postoperative; Recovery Period, Anesthesia
Keywords: Pain Management; Quality of Healthcare
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- serratus anterior plane block (Active Comparator): The serratus anterior plane block will be performed under ultrasound guidance in the preoperative term. Tramadol will be administered via patient controlled analgesia (PCA) device at 20 mg bolus dose with 10 min. lockout time without basal infusion dose.
  Interventions: Procedure: serratus anterior plane block
- erector spina plane block (Active Comparator): The erector spina plane block will be performed under ultrasound guidance in the preoperative term. Tramadol will be administered via PCA device at 20 mg bolus dose with 10 min. lockout time without basal infusion dose.
  Interventions: Procedure: erector spina plane block

INTERVENTIONS:
Procedure: serratus anterior plane block — ultrasound guided serratus anterior plane block will be done with % 0.25 bupivacaine.
  Arms: serratus anterior plane block
Procedure: erector spina plane block — ultrasound guided erector spina plane block will be done with % 0.25 bupivacaine.
  Arms: erector spina plane block

SUMMARY:
The aim of this study is to compare the efficiency of serratus anterior plane block and erector spina plane block on analgesic consumption, postoperative pain and patient's satisfaction and recovery quality in patients undergoing mastectomy.

DETAILED DESCRIPTION:
Mastectomy may cause severe postoperative pain. There are several analgesic methods for postoperative pain management. Serratus anterior plane (SAP) block is an interfascial plane block which is performed into the fascial plane of serratus anterior muscle. It provides effective analgesia in anterior, posterior and lateral dermatomes of thorax. There are several studies about its analgesic efficacy for mastectomy pain. The erector spina plane (ESP) block is another novel plan block which provides analgesia at multi-dermatomal area of the anterior, posterior, and lateral thoracic and abdominal walls. There are some studies about its effectiveness for postoperative mastectomy pain management. However, according to our best knowledge, there is no literature comparing the efficacy of ESP block and SAP block patients undergoing mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* American society of score anesthesiologist I-II-III
* Elective modified radical mastectomy
* 18-65 years old

Exclusion Criteria:

* neurological disease
* coagulopathy disease or using anticoagulants
* non-cooperative
* allergic to one of the drugs used in the study
* recurrent breast cancer
* body mass index is above 35

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-03-18 (Estimated); Primary Completion 2021-02-27 (Estimated); Study Completion 2021-03-15 (Estimated)

PRIMARY OUTCOMES:
Analgesic consumption | From at the end of surgery (at postoperative 0th hour) to postoperative 24th hours
  Tramadol dose will be calculated as milligram

SECONDARY OUTCOMES:
Postoperative pain intensity | At 0,2,4,6,12,24th hours after surgery
  Numeric rating scale which is 0 to 10 will be recorded.In this scale, 0 is no pain, 10 is the worst pain.
Quality of recovery | At postoperative 24th hours
  Quality of recovery (QoR-40) questionaire will be recorded. The QoR-40 is a questionaire which measures of five dimensions of health: patient support, comfort, emotions, physical independence, and pain on a five-point likert scale. QoR-40 scores range from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery)
The number of patients with perioperative side effects | From 30 minute before surgery to postoperative 24th hours
  The number of patients with perioperative side effects(emesis, nausea, local anesthetic toxicity, pneumothorax, local hematoma) will be recorded